CLINICAL TRIAL: NCT06926803
Title: A Clinical Study of Furmonertinib in the Treatment of EGFR-Mutated NSCLC With Leptomeningeal Metastases
Status: Active, not recruiting | Type: Observational
Sponsor: Qiming Wang (Other Government)
Responsible Party: Sponsor-Investigator, Qiming Wang, Director, Henan Cancer Hospital
Organization: Henan Cancer Hospital (Other Government)
Other Study IDs: 2025-019
Record Dates: First submitted 2025-03-05; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-02

CONDITIONS: Lung Cancer (NSCLC); Leptomeningeal Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study adopts a retrospective design. Patients enrolled will include those who received furmonertinib (treatment duration ≥1 month) between March 3, 2021, and December 31, 2024, with concurrent therapies permitted (e.g., radiotherapy, intrathecal chemotherapy, surgical interventions such as ventriculoperitoneal shunting). A retrospective analysis will be conducted to investigate the efficacy and safety of furmonertinib-based therapy (with or without other treatments) in EGFR-mutated NSCLC patients with leptomeningeal metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years, male or female;
2. Histologically or cytologically confirmed diagnosis of **non-small cell lung cancer (NSCLC);
3. " EGFR mutation-positive"(classic or non-classic mutations) confirmed by genetic testing;
4. "Leptomeningeal metastasis" definitively diagnosed by investigators based on "EANO-ESMO diagnostic criteria", involving comprehensive clinical assessment including symptom evaluation, imaging evaluation (MRI/CT), and/or cerebrospinal fluid (CSF) cytology;
5. Received furmonertinib (treatment duration ≥1 month) between "March 3, 2021, and December 31, 2024", with concurrent therapies permitted (e.g., radiotherapy, intrathecal chemotherapy, surgical interventions such as ventriculoperitoneal shunting).

Exclusion Criteria

1. History of other malignancies during NSCLC treatment or prior to diagnosis, except those effectively controlled (e.g., complete remission ≥5 years);
2. Severe gastrointestinal disorders affecting drug administration or absorption, including but not limited to peptic ulcer disease, inflammatory bowel disease, or malabsorption syndromes;
3. Evidence of uncontrolled systemic diseases (e.g., uncontrolled hypertension [BP >140/90 mmHg despite treatment], diabetes mellitus [HbA1c >8%], arrhythmias, heart failure [NYHA class III/IV], active bleeding, active infections requiring IV antibiotics, or interstitial pneumonia requiring corticosteroid therapy), which in the investigator's judgment may directly compromise patient prognosis;
4. Incomplete medical records or follow-up data;
5. Pregnancy or lactation;
6. Other severe acute/chronic medical conditions, psychiatric disorders, or laboratory abnormalities that, in the investigator's opinion, may confound the interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with EGFR-mutated non-small cell lung cancer (NSCLC) and leptomeningeal metastasis who received furmonertinib therapy between **March 3, 2021, and December 31, 2024**, with a treatment duration of ≥1 month.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
OS | The time interval from the first administration of furmonertinib after the diagnosis of leptomeningeal metastasis to the date of death from any cause（up to 60 months））
  overall survival

SECONDARY OUTCOMES:
TTF | Defined as the interval from the first administration of furmonertinib after the diagnosis of leptomeningeal metastasis to the permanent discontinuation of furmonertinib therapy due to disease progression, toxicity, or any other reason（up to 12 months)）
  Time to Treatment Failure
ORR-LM | The proportion of subjects achieving complete response (CR) or partial response (PR) in leptomeningeal lesions, observed from the first administration of furmonertinib after leptomeningeal metastasis diagnosis until disease progression(up to 12 months)
  Objective Response Rate for Leptomeningeal Metastasis

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No